CLINICAL TRIAL: NCT05532241
Title: Environmental Factors and Microbiological Interactions in Structure of Dental Biofilm
Brief Title: Dental Biofilm Control During Orthodontic Treatment
Acronym: ORTHOBIOFILM
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Rijeka (Other)
Collaborators: University of Ljubljana (Other)
Responsible Party: Principal Investigator, Stjepan Spalj, Professor, University of Rijeka
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IP-2020-02-4027
Record Dates: First submitted 2022-05-23; First posted 2022-09-08 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Gingivitis; Malocclusion
Keywords: malocclusion; gingivitis; dental biofilm
MeSH Terms: conditions — Gingivitis; Malocclusion | interventions — Oral Hygiene; Parodontax; halofantrine

STUDY DESIGN:
Intervention Model Description: 2 types of appliances and 2 experimental conditions
Who Masked: Outcomes Assessor
Masking Description: Groups were labeled as I-IV, appliance is fixed on teeth and visible for both participants and care providers. Mouthwash is also visible. Outcome assessor does not know wether patient was in mouthwash group, but he sees the type of appliance. Microbiologist and statisticians are not aware of the group affiliation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- metal + OH (Experimental): fixed metal orthodontic appliance with regular oral hygiene (toothbrush + toothpaste with low concentration of fluorides 1450 ppm)
  Interventions: Device: fixed metal orthodontic appliance; Procedure: oral hygiene
- metal + CHX (Experimental): fixed metal orthodontic appliance with antiseptic mouthwash one-month use (0.12% chlorhexidine digluconate)
  Interventions: Device: fixed metal orthodontic appliance; Drug: Chlorhexidine mouthwash
- non-metal + OH (Placebo Comparator): fixed non-metal orthodontic appliance (ceramic brackets + nylon thread) with regular oral hygiene (toothbrush + toothpaste with low concentration of fluorides 1450 ppm)
  Interventions: Device: fixed non-metal orthodontic appliance; Procedure: oral hygiene
- non-metal + CHX (Active Comparator): fixed non-metal orthodontic appliance (ceramic brackets + nylon thread) with antiseptic mouthwash one-month use (0.12% chlorhexidine digluconate)
  Interventions: Device: fixed non-metal orthodontic appliance; Drug: Chlorhexidine mouthwash

INTERVENTIONS:
Device: fixed metal orthodontic appliance — fixed metal orthodontic appliance (stainless steel brackets (Mini Master MBT 0.022'', American Orthodontics), nickel-titanium archwire (NiTi, American Orthodontics), elastomeric ligatures (Elastomerics, American Orthodontics))
  Other Names: Mini Master MBT 0.022'' and nickel-titanium archwire (American Orthodontics)
  Arms: metal + CHX; metal + OH
Device: fixed non-metal orthodontic appliance — fixed non-metal orthodontic appliance (ceramic brackets (Radiance MBT 0.022'', American Orthodontics), polyamide thread, elastomeric ligatures (Elastomerics, American Orthodontics))
  Other Names: Radiance MBT 0.022'' (American Orthodontics) and polyamide thread
  Arms: non-metal + CHX; non-metal + OH
Procedure: oral hygiene — conducting regular oral hygiene, commonly recommended for orthodontic patients (toothbrush + toothpaste with a low fluoride concentration of 1450 ppm (Parodontax, GSK)
  Other Names: Parodontax (GSK)
  Arms: metal + OH; non-metal + OH
Drug: Chlorhexidine mouthwash — conducting regular oral hygiene (Parodontay, GSK) + 0.12% chlorhexidine digluconate mouthwash (Curasept ADS 212, Curaden) daily during one month
  Other Names: Parodontax (GSK) + Curasept ADS 212 (Curadent)
  Arms: metal + CHX; non-metal + CHX

SUMMARY:
Orthodontic appliances can affect changes in the relationships of members of the oral microbiome. Microbiome imbalance can result in oral infections and complicate treatment. The focus is on the microbiological profile of dental biofilm and its control. The effects of metals released by corrosion of alloys for oral use on the microbiome and the extent to which they modify the effectiveness of gingivitis therapy by mechanical and chemical control of biofilm will be investigated. Early and late colonizers of the tooth surface will be analyzed. The condition of gingiva will be assessed, and the results will show the specifics of biofilm and gingiva exposed and unexposed, and differences in the response of individual bacteria to therapy. Molecular biology techniques will be used to quantify the total bacterial biomass (16s rRNA) and the proportion of specific bacterial species within the dental biofilm.

DETAILED DESCRIPTION:
The aim is:

* to determine the clinical characteristics of gingiva of subjects not exposed to metals of dental alloys and exposed to metals
* characterization of microbiome of dental biofilm in subjects not exposed to metals of dental alloys and exposed to metals and to determine changes in the structure of dental biofilm due to exposure to metals
* examine the extent to which environmental influences modify the effectiveness of treatment of gingivitis by mechanical removal of biofilm and chemical control (chlorhexidine digluconate mouthwash (CHX))
* to examine the behavior of bacteria of early and late colonizers of dental biofilm after chemical control
* to analyze biofilm on metal and non-metal appliance
* to explore patient reported outcome measures Study design is a randomized controlled trial with 4 parallel groups: (I) fixed metal orthodontic appliance with regular oral hygiene, (II) fixed metal orthodontic appliance with CHX, (III) non-metal fixed orthodontic appliance with regular oral hygiene, and (IV) non-metal orthodontic appliance with CHX.

ELIGIBILITY:
Inclusion Criteria:

* malocclusion with moderate or great need for orthodontic treatment (Index of Orthodontic Treatment Need grades >=3)

Exclusion Criteria:

* neurodevelopmental disorders
* intellectual disability
* oligodontia
* congenital craniofacial anomalies
* orofacial clefts

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
bacterial composition of dental biofilm | 90 days (change from start to 2 months and 3 months after start)
  bacterial ratio in dental biofilm (molecular biology analysis)
gingival enlargement | 90 days (change from start to 2 months and 3 months after start)
  Seymour index (thickness (scale 0=normal-2=thickening >=3mm) + proportion of tooth crown coverage (scale 0=normal-3=papilla involving .2/3 of adjacent tooth crown half) on frontal teeth vestibular and oral in both jaws; scale 0-100), higher score means worse outcome

SECONDARY OUTCOMES:
dental biofilm accumulation | 90 days (change from start to 2 months and 3 months after start)
  Silness-Loe index and Williams modification for subjects in orthodontic treatment on a scale from 0=no biofilm to 3=a continuous line greater than 1mm, mean value of referent teeth, range 0-3, higher score indicates worse outcome
pH of biofilm | 90 days (change from start to 2 months and 3 months after start)
  colorimetric test with pH scale in range 4-7, lower score means worse outcome (higher acidity)
extent of gingivitis | 90 days (change from start to 2 months and 3 months after start)
  Full mouth bleeding score on a scale 0-100%, higher score means worse outcome
oral health-related quality of life | 90 days (change from start to 2 months and 3 months after start)
  Oral Health Impact Profile (modification for gingivitis), 8 items, each on a scale 0=never-4=very often, range 0-32, higher score means worse outcome

CONTACTS AND LOCATIONS:
Locations (3):
- Croatia (3):
  - University of Rijeka Faculty of Dental Medicine, Rijeka
  - University of Rijeka, Faculty od Dental Medicine, Dental Clinic, Rijeka
  - University of Rijeka, Faculty of Dental Medicine, Rijeka

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be shared on reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: March 2024
Access Criteria: No criteria established

REFERENCES:
- See also: This research is a part of a larger project described on this site — https://sites.google.com/view/ip-2020-02/početna-stranica